CLINICAL TRIAL: NCT00869817
Title: Dominantly Inherited Alzheimer Network (DIAN)
Acronym: DIAN
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IA0147; U19AG032438 (NIH)
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; antecedent biomarkers; Amyloid Precursor Protein (APP) mutation; presenilin I (PS1) mutation; presenilin 2 (PS2) mutation; Autosomal Dominant Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Alzheimer disease, familial, type 3; Alzheimer disease type 4

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — buffy coat, plasma, cerebral spinal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Mutation Positive
- 2: Mutation Negative

SUMMARY:
The purpose of this study is to identify potential biomarkers that may predict the development of Alzheimer's disease in people who carry an Alzheimer's mutation.

DETAILED DESCRIPTION:
Dominantly inherited Alzheimer's disease (AD) represents less than 1% of all cases of AD and is an important model for study because the responsible mutations have known biochemical consequences that are believed to underlie the pathological basis of the disorder. Three major hypotheses will be tested:

* First, that there is a period of preclinical (presymptomatic) AD in individuals who are destined to develop early-onset dementia (gene carriers) that can be detected by changes in biological fluids and in neuroimaging correlates in comparison with individuals who will not develop early-onset dementia (non-carriers).
* Second, because all identified causative mutations for AD affect the normal processing of amyloid precursor protein (APP) and increase brain levels of amyloid-beta 42 (Aβ42), the sequence of preclinical changes initially will involve Aβ42 (production and clearance; reduced levels in cerebrospinal fluid [CSF]), followed by evidence for cerebral deposition of Aβ42 (amyloid imaging), followed by cerebral metabolic activity (functional imaging), and finally by regional atrophy (structural imaging).
* Finally, that the phenotype of symptomatic early-onset familial AD, including its clinical course, is similar to that of late-onset "sporadic" AD.

The following specific aims will be used to test these hypotheses:

1. Maintain the established international DIAN registry of individuals (MCs and non-carriers (NC), symptomatic and asymptomatic) who are biological adult children of an affected parent with an APP, PSEN1, or PSEN2 mutation causing AD and assess participants every 2 years with the uniform DIAN protocol.
2. Recruit to the registry 50 new asymptomatic participants, both MCs and NCs, in Year 1 of the next budget period to maintain the total DIAN cohort at ~250 individuals. These new participants will include those who are more than 15 years younger than the estimated age of symptomatic onset (EAO) to explore the earliest observable biomarker changes of preclinical AD.
3. Maintain the integrated DIAN database and biospecimen repository to disseminate data and tissue to qualified investigators (within and outside of DIAN) in a user-friendly manner and to permit analyses within, between, and among the various data domains that will include:

   1. In asymptomatic MCs (using NCs as controls), determine the temporal ordering and rate of intraindividual change in clinical, cognitive, imaging, and fluid biomarkers of AD prior to EAO
   2. In symptomatic MCs, compare the clinical and neuropathological phenotypes of ADAD to those of LOAD, using datasets such as ADNI.
4. Utilize the DIAN cohort and its database and biospecimen repository to support new scientific studies, including use of exome chip technology to examine potential modifiers of age at symptomatic onset. Pursue other new scientific initiatives that are funded independently of the DIAN grant but are conducted within the DIAN infrastructure at no cost to DIAN including: Dermal fibroblasts and induced pluripotent stem cells (iPSCs), examine biomarker surrogates for neurogeneration in CSF including Visinin-like protein-1 (VILIP-1), Tau seeding assay, Stable Isotope Leucine Kinetics (SILK) in DIAN participants, determine the exact Abeta species that underlie AD pathology using Mass spectrometry, exome sequencing on all DIAN participants to search for both positive and negative modifiers of EYO, and amyloid imaging crossover to [18F]florbetapir.
5. Provide genetic counseling to any and all DIAN participants who wish to learn their mutation status and, for those who decide to learn their status after counseling, provide genetic testing by Clinical Laboratory Improvement Amendments (CLIA)-approved laboratories (i.e., outside of DIAN).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from participant and collateral source prior to any study-related procedures.
* Aged 18 (inclusive) or older and the child of an affected individual (clinically or by testing) in a pedigree with a known mutation for ADAD.
* Cognitively normal to very mild or mild cognitive impairment (CDR score range 0-1.0). Primary enrollment will focus on the recruitment of asymptomatic adult children who are more than 15 years younger than the estimated age of symptom onset. Enrollment of new participants with moderate cognitive impairment is allowed with the prior approval of the DIAN Coordinating Center.
* Has two persons who are not their full-blooded siblings who can serve as collateral sources for the study.
* Fluent in a language approved by the DIAN Coordinating Center at about the 6th grade level (international equivalent) or above.

Exclusion Criteria:

* Under age 18
* Medical or psychiatric illness that would interfere in completing initial and follow-up visits
* Requires nursing home level care
* Has no one who can serve as a study informant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mutation carriers and non-carriers from families with a mutation (which is different from the genetic risk factor Apo-E4) known to cause Alzheimer's disease.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2009-01; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Positive predictive power of a biomarker or group of biomarkers | Variable follow-up assessment based on age in relation to age at onset of affected parent.
Biomarkers obtained by blood draw, lumbar puncture, MRI, FDG PET, PET amyloid imaging | Variable follow-up assessment based on age in relation to age at onset of affected parent
Clinical markers also examined from clinical interview and cognitive testing | Variable follow-up assessment based on age in relation to age at onset of affected parent

CONTACTS AND LOCATIONS:
Overall Officials: Eric McDade, DO, Principal Investigator — Washington University School of Medicine; Alisha Daniels, MD,MHA, Study Director — (314) 273-9057
Locations (26):
- United States (8):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Indiana University-Indiana Alzheimer Disease Center, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Columbia University, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - University of Washington, Seattle, Washington
- Argentina (2):
  - Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia" (FLENI) Instituto de Investigaciones Neurológicas Raúl Correa, Buenos Aires
  - Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia (FLENI), Salta
- Australia (3):
  - Neuroscience Research Australia, Sydney, New South Wales
  - Mental Health Research Institute, University of Melbourne, Melbourne, Victoria
  - Sir James McCusker Alzheimer's Disease Research Unit, Edith Cowan University, Perth, Western Australia
- Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil
- McGill University Research Centre for Studies in Aging, Verdun, Quebec, Canada
- Grupo Neurociencias de Antioquia, Medellín, Colombia
- Germany (2):
  - German Center for Neurodegenerative Diseases (DZNE) Munich, and University Hospital Ludwig-Maximilians-Universitat (LMU) Munich, Munich
  - German Center for Neurodegenerative Diseases (DZNE) Tübingen and Hertie-Institute for Clinical Brain Research, University of Tübingen, Tübingen
- Japan (3):
  - Niigata University, Niigata
  - Osaka City University, Osaka
  - Tokyo University, Tokyo
- Instituto Nacional de Neurología y Neurocirugía "Manuel Velasco Suarez", Mexico City, Mexico
- Amsterdam UMC, Amsterdam, Netherlands
- Asan Medical Center, Seoul, Songpa-Gu, South Korea
- Hospital Clinic Barcelona, Barcelona, Catalonia, Spain
- Institute of Neurology, Queen Square, London, United Kingdom

REFERENCES:
- [Background] Mintun MA, Larossa GN, Sheline YI, Dence CS, Lee SY, Mach RH, Klunk WE, Mathis CA, DeKosky ST, Morris JC. [11C]PIB in a nondemented population: potential antecedent marker of Alzheimer disease. Neurology. 2006 Aug 8;67(3):446-52. doi: 10.1212/01.wnl.0000228230.26044.a4. PMID 16894106
- [Background] Fagan AM, Roe CM, Xiong C, Mintun MA, Morris JC, Holtzman DM. Cerebrospinal fluid tau/beta-amyloid(42) ratio as a prediction of cognitive decline in nondemented older adults. Arch Neurol. 2007 Mar;64(3):343-9. doi: 10.1001/archneur.64.3.noc60123. Epub 2007 Jan 8. PMID 17210801
- [Background] Godbolt AK, Cipolotti L, Anderson VM, Archer H, Janssen JC, Price S, Rossor MN, Fox NC. A decade of pre-diagnostic assessment in a case of familial Alzheimer's disease: tracking progression from asymptomatic to MCI and dementia. Neurocase. 2005 Feb;11(1):56-64. doi: 10.1080/13554790490896866. PMID 15804925
- [Background] Morris JC, McKeel DW Jr, Storandt M, Rubin EH, Price JL, Grant EA, Ball MJ, Berg L. Very mild Alzheimer's disease: informant-based clinical, psychometric, and pathologic distinction from normal aging. Neurology. 1991 Apr;41(4):469-78. doi: 10.1212/wnl.41.4.469. PMID 2011242
- [Background] Galvin JE, Powlishta KK, Wilkins K, McKeel DW Jr, Xiong C, Grant E, Storandt M, Morris JC. Predictors of preclinical Alzheimer disease and dementia: a clinicopathologic study. Arch Neurol. 2005 May;62(5):758-65. doi: 10.1001/archneur.62.5.758. PMID 15883263
- [Derived] Wagemann O, Li Y, Hassenstab J, Aschenbrenner AJ, McKay NS, Gordon BA, Benzinger TLS, Xiong C, Cruchaga C, Renton AE, Perrin RJ, Berman SB, Chhatwal JP, Farlow MR, Day GS, Ikeuchi T, Jucker M, Lopera F, Mori H, Noble JM, Sanchez-Valle R, Schofield PR, Morris JC, Daniels A, Levin J, Bateman RJ, McDade E, Llibre-Guerra JJ; Dominantly Inherited Alzheimer Network. Investigation of sex differences in mutation carriers of the Dominantly Inherited Alzheimer Network. Alzheimers Dement. 2024 Jan;20(1):47-62. doi: 10.1002/alz.13460. Epub 2023 Sep 23. PMID 37740921
- [Derived] Prescott JW, Doraiswamy PM, Gamberger D, Benzinger T, Petrella JR; Dominantly Inherited Alzheimer Network. Diffusion Tensor MRI Structural Connectivity and PET Amyloid Burden in Preclinical Autosomal Dominant Alzheimer Disease: The DIAN Cohort. Radiology. 2022 Jan;302(1):143-150. doi: 10.1148/radiol.2021210383. Epub 2021 Oct 12. PMID 34636637
- [Derived] Gordon BA, Blazey TM, Su Y, Hari-Raj A, Dincer A, Flores S, Christensen J, McDade E, Wang G, Xiong C, Cairns NJ, Hassenstab J, Marcus DS, Fagan AM, Jack CR Jr, Hornbeck RC, Paumier KL, Ances BM, Berman SB, Brickman AM, Cash DM, Chhatwal JP, Correia S, Forster S, Fox NC, Graff-Radford NR, la Fougere C, Levin J, Masters CL, Rossor MN, Salloway S, Saykin AJ, Schofield PR, Thompson PM, Weiner MM, Holtzman DM, Raichle ME, Morris JC, Bateman RJ, Benzinger TLS. Spatial patterns of neuroimaging biomarker change in individuals from families with autosomal dominant Alzheimer's disease: a longitudinal study. Lancet Neurol. 2018 Mar;17(3):241-250. doi: 10.1016/S1474-4422(18)30028-0. Epub 2018 Feb 1. PMID 29397305
- [Derived] Bateman RJ, Xiong C, Benzinger TL, Fagan AM, Goate A, Fox NC, Marcus DS, Cairns NJ, Xie X, Blazey TM, Holtzman DM, Santacruz A, Buckles V, Oliver A, Moulder K, Aisen PS, Ghetti B, Klunk WE, McDade E, Martins RN, Masters CL, Mayeux R, Ringman JM, Rossor MN, Schofield PR, Sperling RA, Salloway S, Morris JC; Dominantly Inherited Alzheimer Network. Clinical and biomarker changes in dominantly inherited Alzheimer's disease. N Engl J Med. 2012 Aug 30;367(9):795-804. doi: 10.1056/NEJMoa1202753. Epub 2012 Jul 11. PMID 22784036
- See also: DIAN Website — https://dian.wustl.edu/
- See also: Washington University St. Louis Knight Alzheimer's Disease Research Center — http://knightadrc.wustl.edu/